CLINICAL TRIAL: NCT02999841
Title: Effect of Acarbose and Vildagliptin on Visceral Fat Distribution in Overweight and Obesity Patients With Newly Diagnosed Type 2 Diabetes Mellitus: A Randomized Control Study
Brief Title: Effect of Acarbose and Vildagliptin on Visceral Fat Distribution in Newly Diagnosed Type 2 Diabetes Patients
Acronym: VISA-T2DM
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Linong Ji, Director of Department of Endocrinology and Metabolism, Peking University People's Hospital., Peking University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2119000273
Record Dates: First submitted 2016-03-15; First posted 2016-12-21 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-12

CONDITIONS: Diabetes Mellitus, Type 2; Obesity
Keywords: Visceral fat
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Acarbose; Vildagliptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Acarbose
  Interventions: Drug: Acarbose
- Group B (Active Comparator): Vildagliptin
  Interventions: Drug: Vildagliptin

INTERVENTIONS:
Drug: Acarbose — 1-2 week: 50mg tid; 3-24 week: 100mg tid.
  Other Names: Glucobay (Acarbose Tablets)
  Arms: Group A
Drug: Vildagliptin — 1-24 week: 50mg bid
  Other Names: Galvus (Vidagliptin Tablets)
  Arms: Group B

SUMMARY:
Focusing on newly diagnosed type 2 diabetes participants with overweight and obesity (24kg/m2 ≤ body mass index ≤ 30kg/m2).

50 participants per arm (acarbose & lifestyle combination / vildagliptin & lifestyle combination), using abdominal computed tomography scans and other methods to evaluate the effects of acarbose and vildagliptin on visceral fat distribution in overweight and obesity patients with newly diagnosed type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* All patients was diagnosed within the past 12 months with type 2 diabetes patients (WHO, 1999 criteria ).
* Not received oral anti-diabetic drugs or has been on short-term(1month) treatment that had been discontinued 3 months before enrollment.
* 30 ≤ Age ≤ 70 years old, male or female.
* HbA1c between 7% and 9% (7.0% ≤ HbA1c ≤9.0%).
* 24 ≤ BMI ≤ 30 kg/m2.
* Written Informed consent.

Exclusion Criteria:

* Subject with type 1 diabetes or gestational diabetes mellitus and other specific types DM.
* Those who can not tolerate AGI or who is suffering GI disease.
* Subject with repeated severe hypoglycemia and/or unawareness of hypoglycemia.
* Known or suspected allergy to trial product(s) or related products.
* Females of child bearing potential who are pregnant, breast-feeding or have the intention of becoming pregnant or not using adequate contraceptive methods throughout the trial
* Impaired liver function, defined as ALT≥2 or AST≥ 2 times upper referenced limit times upper normal limit.
* Any other clinically significant condition or major systemic diseases, including serious coronary heart disease, cardiovascular disease, cancer, TB, acute infection.
* Endocrine diseases (hypo thyroidism, hyperthyroidism,Cushing's syndrome).
* Uncontrolled hypertension(SBP≥180mmHg and/or DBP≥100mmHg).
* Diabetic ketoacidosis; or hyperosmolar non-ketotic coma.
* Concomitant treatment which influences blood glucose and bodyweight.
* Impaired renal function(Cr≥ 1.5 mg/dl in male or Cr≥1.4 mg/dl in female).
* Mental disorders; drug or other substance misuse.
* Participation in any drug clinical trials during the past 3 months before enrolment.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-12 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Change of the visceral fat area in square centimeter assessed by abdominal CT scans from baseline to 24 weeks. | 24 weeks

SECONDARY OUTCOMES:
Change of body weight in kilograms measured by investigators from baseline to 24 weeks. | 24 weeks
Change of waist circumstance in centimeters measured by investigators from baseline to 24 weeks. | 24 weeks
Change of body mass index in kg/m^2 measured by investigators from baseline to 24 weeks. | 24 weeks
Change of the subcutaneous fat area in square centimeters assessed by abdominal CT scans from baseline to 24 weeks. | 24 weeks
Change of hemoglobin A1c in percents from baseline to 24 weeks. | 24 weeks
Change of hemoglobin fasting plasma glucose in millimols per liter from baseline to 24 weeks. | 24 weeks
Change of hemoglobin 2-hour-post-prandial plasma glucose in millimols per liter from baseline to 24 weeks. | 24 weeks
Change of triglyceride in millimols per liter from baseline to 24 weeks. | 24 weeks
Change of total cholesterol in millimols per liter from baseline to 24 weeks. | 24 weeks
Change of low-density lipoprotein-cholesterol in millimols per liter from baseline to 24 weeks. | 24 weeks
Change of high-density lipoprotein-cholesterol in millimols per liter from baseline to 24 weeks. | 24 weeks
Change of insulin in international units per liter from baseline to 24 weeks. | 24 weeks
Change of brain natriuretic peptide in nanograms per milliliter from baseline to 24 weeks. | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Linong Ji, MD, Principal Investigator — Peking University People's Hospital
Locations (1):
- Beijing Pinggu Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Do not share data.

REFERENCES:
- [Result] Ibrahim MM. Subcutaneous and visceral adipose tissue: structural and functional differences. Obes Rev. 2010 Jan;11(1):11-8. doi: 10.1111/j.1467-789X.2009.00623.x. Epub 2009 Jul 28. PMID 19656312
- [Result] Schernthaner GH, Schernthaner G. Insulin resistance and inflammation in the early phase of type 2 diabetes: potential for therapeutic intervention. Scand J Clin Lab Invest Suppl. 2005;240:30-40. doi: 10.1080/00365510500236119. PMID 16112958
- [Result] Monami M, Iacomelli I, Marchionni N, Mannucci E. Dipeptydil peptidase-4 inhibitors in type 2 diabetes: a meta-analysis of randomized clinical trials. Nutr Metab Cardiovasc Dis. 2010 May;20(4):224-35. doi: 10.1016/j.numecd.2009.03.015. Epub 2009 Jun 9. PMID 19515542
- [Result] Kodama N, Tahara N, Tahara A, Honda A, Nitta Y, Mizoguchi M, Kaida H, Ishibashi M, Abe T, Ikeda H, Narula J, Fukumoto Y, Yamagishi S, Imaizumi T. Effects of pioglitazone on visceral fat metabolic activity in impaired glucose tolerance or type 2 diabetes mellitus. J Clin Endocrinol Metab. 2013 Nov;98(11):4438-45. doi: 10.1210/jc.2013-2920. Epub 2013 Sep 12. PMID 24030946
- [Derived] Yang X, Zhang X, Sun C, Zhao C, Kong X, Zhao M, Ji L, Li Y. Effect of acarbose and vildagliptin on plasma trimethylamine N-oxide levels in patients with type 2 diabetes mellitus: a 6-month, two-arm randomized controlled trial. Front Endocrinol (Lausanne). 2025 May 6;16:1575087. doi: 10.3389/fendo.2025.1575087. eCollection 2025. PMID 40395816
- [Derived] Zhang X, Ren H, Zhao C, Shi Z, Qiu L, Yang F, Zhou X, Han X, Wu K, Zhong H, Li Y, Li J, Ji L. Metagenomic analysis reveals crosstalk between gut microbiota and glucose-lowering drugs targeting the gastrointestinal tract in Chinese patients with type 2 diabetes: a 6 month, two-arm randomised trial. Diabetologia. 2022 Oct;65(10):1613-1626. doi: 10.1007/s00125-022-05768-5. Epub 2022 Aug 5. PMID 35930018